CLINICAL TRIAL: NCT03141021
Title: Multi-Institutional Registry for Malignant Peripheral Nerve Sheath Tumors
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Boston's Children Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201702006
Record Dates: First submitted 2017-04-13; First posted 2017-05-04 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Malignant Peripheral Nerve Sheath Tumors
MeSH Terms: conditions — Neurofibrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Biospecimens collected under associated banks (frozen or paraffin-embedded, germline (or normal tissue DNA) samples, and any previously somatic whole-exome or whole-genome sequencing data for aggregate analyses) and prospectively collect MPNST samples for analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
First, the investigators plan to use a retrospective analysis to determine the clinical landscape of neurofibromatosis (NF)1-associated malignant peripheral nerve sheath tumor (MPNST) and precursor lesions (e.g., atypical or nodular plexiform neurofibromas). A worldwide database will be established, collecting, in a standardized manner, histologic, immunohistochemical, molecular, radiographic, treatment, and related clinical data from centers worldwide with expertise in these NF1-related cancers. Although retrospective in nature, the resulting data from this registry may reveal previously unanticipated patterns, similar to the INFACT effort outcome. This registry would then allow the acquisition of data associated with MPNST biospecimens collected under associated banks (frozen or paraffin-embedded, germline (or normal tissue DNA) samples, and any previously somatic whole-exome or whole-genome sequencing data for aggregate analyses). Second, the investigators plan to co-register patients to institutional banks in order to prospectively collect MPNST samples for analysis. These patients will be consented in order to collect the above information and for banking of tumor tissue and future studies that include genomic characterization of the tumors.

ELIGIBILITY:
Inclusion Criteria and Exclusion Criteria:

-Any patient diagnosed with an MPNST is eligible for enrollment to this registry provided s/he consents to participate (or consent form his/her parent or legal guardian or legally authorized representative is obtained).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The oncology clinic of each participating institution
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2053-04-30 (Estimated); Study Completion 2053-04-30 (Estimated)

PRIMARY OUTCOMES:
Histologic characteristics of malignant peripheral nerve sheath tumor (MPNST) | 10 years
  -The data collected through this registry will be used to analyze previously unanticipated patterns and prognostic clues about MPNST
Immunohistochemical characteristics of malignant peripheral nerve sheath tumor (MPNST) | 10 years
  -The data collected through this registry will be used to analyze previously unanticipated patterns and prognostic clues about MPNST
Molecular characteristics of malignant peripheral nerve sheath tumor (MPNST) | 10 years
  -The data collected through this registry will be used to analyze previously unanticipated patterns and prognostic clues about MPNST
Radiographic characteristics of malignant peripheral nerve sheath tumor (MPNST) | 10 years
  -The data collected through this registry will be used to analyze previously unanticipated patterns and prognostic clues about MPNST
Treatment given to patients with malignant peripheral nerve sheath tumor (MPNST) | 10 years
  -The data collected through this registry will be used to analyze previously unanticipated patterns and prognostic clues about MPNST
Future genomic characterization of malignant peripheral nerve sheath tumor (MPNST) | 10 years
  -The data collected through this registry will be used to analyze previously unanticipated patterns and prognostic clues about MPNST

CONTACTS AND LOCATIONS:
Overall Officials: Angela Hirbe, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (13):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins, Baltimore, Maryland
  - National Institutes of Health (NIH), Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Lifespan, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah
- Mount Sinai, Toronto, Ontario, Canada
- Global Gene Corporation, Mumbai, India
- Nagoya University Hospital, Nagoya, Showa Ward, Japan
- Royal National Orthopedic Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu